CLINICAL TRIAL: NCT04047745
Title: The Use of Liposomal Bupivacaine Interscalene Brachial Plexus Block for Rotator Cuff Surgery: A Randomized, Double Blind, Clinical Trial
Brief Title: Post-operative Exparel Study Following Rotator Cuff Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019Tucker
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liposomal bupivacaine (Active Comparator)
  Interventions: Drug: Liposomal bupivacaine
- ropivacaine (Active Comparator)
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Liposomal bupivacaine — interscalene nerve block administered before surgery using 133 mg liposomal bupivacaine with 10mL 0.5% ropivacaine
  Arms: liposomal bupivacaine
Drug: Ropivacaine injection — interscale nerve block administered before surgery using 30mL 0.5% ropivacaine
  Arms: ropivacaine

SUMMARY:
The primary purpose of this study is to determine if the postoperative oral narcotics consumption in patients receiving liposomal bupivacaine (LB) interscalene brachial plexus nerve block (ISBPB) is different than the narcotics consumption receiving traditional bupivacaine ISBPB for arthroscopic rotator cuff repair analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 years or older with a full-thickness rotator cuff tear (confirmed on MRI) undergoing arthroscopic rotator cuff repair surgery.
* Anesthesiologists physical status 1, 2, or 3 and normal preoperative motor (Lovett scale: biceps, wrist, thumb) and sensory function.

Exclusion Criteria:

* Revision shoulder surgery
* History of more than 1 prior surgery performed on the operative shoulder
* Concomitant severe glenohumeral arthritis
* Concomitant adhesive capsulitis
* Worker's compensation claim
* Pregnancy
* History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics
* History of renal or hepatic failure
* Chronic neuromuscular deficit affecting the surgical limb.
* Uncontrolled psychiatric or neurologic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
opioid consumption | surgery through 48 hours post-op
  postsurgical opioid consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedics at Egg Harbor Township, Egg Harbor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No